CLINICAL TRIAL: NCT04280094
Title: Can the Ideal Mesh Size be Standardized for Open Inguinal Hernia Repair; An Anthropometric Study in Central Anatolian Male Patients
Brief Title: Can Ideal Mesh Size be Standardized in Open Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, principal investigator, Konya Meram State Hospital
Other Study IDs: SBU Konya SUAM
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Two hundred consecutive unilateral inguinal hernia patients will be included in the study. Patients will be recorded by measuring the distance between the pubic tubercle and the deep inguinal ring, the distance between the inguinal ligament and the internal oblique aponeurosis, the distance between the deep and superficial inguinal ring diameters and their anterior superior iliac spine. The contribution of these measures to the determination of the ideal mesh size will be analyzed.

DETAILED DESCRIPTION:
This prospective study includes 200 consecutive male patients who underwent unilateral open inguinal hernia repair since March 2020. Under-18 hernias, complicated hernias, recurrent hernias, and those with laparoscopic hernia repair will be excluded. Initially, the distance between the pubic tubercle and the medial edge of the deep inguinal ring will be measured. Next, the distance between the inner edge of the inguinal ligament and the upper level of the internal oblique aponeurosis will be measured at the Hesselbach triangle. Hesselbach triangle area will be calculated. The diameter of the superficial and deep inguinal ring and their spina iliaca anterior superior (SIAS) distance will be measured. The contribution of these measures to the determination of the ideal mesh size will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male patients over 18 years of age who applied for inguinal hernia surgery

Exclusion Criteria:

* Patients under the age of 18
* Complicated hernias
* Recurrent hernias
* Those undergoing laparoscopic hernia repair

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male patients over the age of 18 who apply to the hospital for inguinal hernia surgery constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Can Ideal Mesh Size be Standardized in Open Inguinal Hernia Repair | The time period of the study was determined as 1 March 2020 and 15 May 2020.
  Patients will be recorded by measuring the distance between the pubic tubercle and the deep inguinal ring, the distance between the inguinal ligament and the internal oblique aponeurosis, the distances between the deep and superficial inguinal ring diameters and the anterior superior iliac spine. Then the data will be analyzed in the SPSS statistics program. Average, maximum, and minimum values of anatomical dimensions will be subtracted. Relationships with age, body length, and body mass index will be analyzed statistically, and the ideal mesh size detectability will be investigated. When the analysis is completed, the study will be terminated.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to share if it is not necessary

REFERENCES:
- [Background] Kulacoglu H, Celasin H, Oztuna D. Individual mesh size for open anterior inguinal hernia repair: an anthropometric study in Turkish male patients. Hernia. 2019 Dec;23(6):1229-1235. doi: 10.1007/s10029-019-01993-x. Epub 2019 Jun 20. PMID 31222460
- [Background] Anitha B, Aravindhan K, Sureshkumar S, Ali MS, Vijayakumar C, Palanivel C. The Ideal Size of Mesh for Open Inguinal Hernia Repair: A Morphometric Study in Patients with Inguinal Hernia. Cureus. 2018 May 3;10(5):e2573. doi: 10.7759/cureus.2573. PMID 29974028